CLINICAL TRIAL: NCT06062693
Title: New Interactive Sensor-home-based Hand Training to Improve Dexterity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02300
Record Dates: First submitted 2023-09-04; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Multiple Sclerosis; Parkinson Disease
Keywords: dexterity; training
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: sensor-home-based hand training for MS, PD, stroke or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- smart sensor egg training (Experimental): An interactive hand trainer with integrated sensors was developed and can be used as input devices to a training which runs on the smartphone or tablet computer to train different finger, hand, and wrist functions.
  Interventions: Device: smart sensor egg training

INTERVENTIONS:
Device: smart sensor egg training — The portable hand trainer has three principal functionalities: (I) Grasping, (II) Pronosupination, and (III) wrist and finger extension. Different exercises can be done.

SUMMARY:
Primary objective of this study is to explore the impact of a 3-week upper limb hand function training in patients with PD, MS or stroke. The benefits on hand function of this training program will be evaluated. The hypothesize is that the 3-week upper limb hand function training improves finger dexterity.

DETAILED DESCRIPTION:
Patients with Parkinson's disease (PD), multiple sclerosis (MS) or stroke often suffer from significantly decreased coordination and have difficulties with precise hand/finger movements during the performance of both basic activities of daily living (ADL), such as dressing, grooming as well as higher ADL, such as cooking, shopping and regular medication intake. The investigators explore the effects of a new, interactive, sensor-home-based upper limb hand training on upper limb related ADL in patients with PD, MS or stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed PD, according to UK Brain bank Criteria (Hughes et al., 1992) or
* MS patients with relapsing-remitting MS (RRMS), secondary-progressive MS (SPMS) or primary progressive MS (PPMS) according to the revised McDonald's criteria or
* subacute stroke
* written and signed informed consent
* self-reported hand function problems

or

* healthy subject
* written and signed informed consent
* no self-reported hand function problems

Exclusion Criteria:

* MoCA <21/30
* psychiatric disease
* participation on other interventional trials
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
hand dexterity | 3 weeks
  Nine Hole Peg test (9-HPT): The 9-HPT is a standardized, well established, and reliable measure of hand dexterity in patients with PD, MS, or stroke. seconds will be measured.

SECONDARY OUTCOMES:
fine finger movements | 3 weeks
  Coin rotation task (CRT): The CRT measures fine coordinated finger movements and is a suitable and valid dexterity test in patients with PD, MS, or stroke. The seconds for 20 halfturns will be measured.
grip strength | 3 weeks
  The handheld JAMAR dynamometer measures the grip strength. kg will be measured.
cognition | baseline
  Montreal Cognitive Assessment (MOCA): Cognitive screening tool with a scale from 0 - 30 points. A higher score means a better outcome.
executive function | 3 weeks
  Trail Making Tests (TMT) parts A & B. Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
executive function | 3 weeks
  Stroop-test: Results are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
self-reported dexterity related problems in daily living for PD | 3 weeks
  Patients with PD: Dexterity Questionnaire 24 (DextQ-24): This questionnaire is a standardized patient self-rated outcome measure (PROM) for evaluating dexterity related ADL in PD. score range 24-96, higher scores mean more dexterity problems.
self-reported arm and hand function related problems in patients with MS | 3 weeks
  Patients with MS: The Arm Function in Multiple Sclerosis Questionnaire (AMSQ): This questionnaire is a standardized patient self-rated outcome measure (PROM) for evaluating arm and hand function in patients with MS. Containing 31 items with a range of 1 - 100 points. Higher scores indicate more limitations in hand and arm function.
Arm and hand function in stroke patients | 3 weeks
  Patients with stroke: Upper limb limos: Mesures arm and hand function in ADL.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanbellingen, Prof. Dr. phil., Principal Investigator — Luzerner Kantonsspital, Universität Bern
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No